CLINICAL TRIAL: NCT04367246
Title: Clinical and Molecular Studies of Li-Fraumeni Syndrome and TP53-associated Disorders
Brief Title: Li-Fraumeni Syndrome/TP53 Biobank
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Kara Maxwell, MD, PhD, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 24919; IRB 18-015810 (Other: Children's Hospital of Philadelphia); IRB 834147 (Other: University of Pennsylvania)
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Li-Fraumeni Syndrome; Li-Fraumeni-Like Syndrome
Keywords: TP53; TP53 Mutation
MeSH Terms: conditions — Li-Fraumeni Syndrome; Li-Fraumeni-Like Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — For affected patients (group 1), collection of biospecimens will occur either once (i.e., blood, buccal swabs, urine, skin fibroblasts), or every six months (i.e., plasma from blood, stool samples, and other specimens that are obtained and leftover as part of clinical care) . Unaffected family members (group 2) and household members (group 3) will only have samples requested once as per Schedule of Study Procedures (Group 3 subjects will not be asked for a germline specimen). None of these procedures are required for the subjects to participate in the study. Children <18 years will complete procedures at CHOP, and adult participants will complete study procedures at PENN (adolescents and young adults seen at CHOP clinically may have their samples collected at CHOP even if over 18 years).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Affected Patients: Eligible subjects have a confirmed germline TP53 mutation or variant, OR have a family history of LFS and clinically managed as a LFS patient, OR meet LFS diagnostic criteria including Classic, Chompret, and LFL (Birch and Eeles) criteria. Medical information contribution is required for participation in the study. Subjects also have options to contribute a one-time DNA sample, a blood sample for plasma and a stool sample every six months, as well as access to their residual clinical tissues.
  Interventions: Other: No Intervention
- Family Members: Biological relative of subjects with germline TP53 mutation or variant (LFS), including first degree (siblings, parents) and second degree (grandparents, aunts, uncles) relatives. Negative for germline TP53 mutation or variant. Medical information contribution is required for participation in the study. Subjects also have options to contribute a one-time DNA sample, a stool sample, as well as access to their residual clinical tissues.
  Interventions: Other: No Intervention
- Household Members: Household member of subjects with germline TP53 mutation or variant (LFS), sharing a living space (apartment or free-standing home) for at least 6 months prior to study enrollment. Medical information contribution is required for participation in the study. Subjects also have options to contribute a one-time stool sample.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention is assigned.

SUMMARY:
Li-Fraumeni Syndrome (LFS) and Li-Fraumeni-like (LFL) Syndrome are cancer predisposition syndromes due to germline aberrations in the TP53 gene. Patients with classical LFS have a lifetime malignancy risk between 80-90%, with 21% of those cancers occurring by the age of 15 years. There are established guidelines for screening patients with LFS that have led to earlier detection and treatment of cancer in this population. There are a number of important issues facing patients identified to have germline TP53 variations. First, with the advent of massively parallel sequencing, increasing numbers of patients are now being identified with a wide range of clinical phenotypes associated with germline TP53 mutations, and the natural history of these patients is less well understood. Second, surveillance for malignancy in LFS and other TP53-associated syndromes involves frequent laboratory and radiologic studies that are imperfect measures of disease onset; therefore, more specific, less invasive biomarker-driven screening methods are needed. Finally, studies to date have not yet identified whether tumors which form in LFS or other germline TP53-associated tumors have unique aberrations or signatures that could be exploited in precision medicine treatment of these patients. In order to study these important issues in LFS, this protocol will establish a TP53 Clinical Database and Biobank. The Investigator plans to use this biobank to study genotype-phenotype correlations in patients with LFS and other germline TP53-associated syndromes, mechanisms of tumor formation, and novel methods of cancer screening in this high risk population.

DETAILED DESCRIPTION:
Context: Li-Fraumeni Syndrome (LFS) and Li-Fraumeni-like (LFL) Syndrome are cancer predisposition syndromes due to germline aberrations in the TP53 gene. Patients with classical LFS have a lifetime malignancy risk between 80-90%. There are guidelines for screening patients with LFS that have led to earlier detection and treatment of cancer in this population. There are a number of important issues facing patients identified to have germline TP53 variations, including study of genotype-phenotype correlations, enhanced cancer screening modalities, and novel treatment strategies for cancers that develop.

Objectives: In order to study important clinical issues in LFS, the primary objective of this biobank is to gather and store ongoing clinical data and biospecimens from patients with LFS and other potential germline TP53-associated syndromes. The investigators plan to use this biobank to study genotype-phenotype correlations in patients with inherited TP53 mutations, mechanisms of tumor formation, and methods of cancer screening.

Study Design: This study is a retrospective/prospective biobank containing clinical data and data and biospecimen. Patients for inclusion will be identified by query of our clinical electronic medical record from the Children's Hospital of Philadelphia (CHOP) and Penn Medicine (PENN) for patients followed in our respective clinics. In addition, patients will be recruited by ongoing prospective collection in clinic. Data collection, data entry and biobank maintenance, will be conducted by the investigators listed on this protocol at CHOP and at PENN through the Master Reliance Agreement. Future investigators and collaborators at other institutions will have access to samples and limited data by executing a written Data User Agreement and/or Materials Transfer Agreement with the biobank.

Setting/Participants: The biobank will be conducted at CHOP and PENN. Any infant, child, or adult with a germline TP53 mutation will be invited to participate. In addition, individuals with a diagnosis of LFS or LFL, who have been seen by a physician at Penn/CHOP or referred from outside physicians will be contacted for participation. To provide control group samples, unaffected family members and/or household members will also be recruited. Prospective enrollment into the biobank is planned to be an ongoing effort, without a fixed end date or target subject number. At minimum, however, the estimated number of recruitment is approximately 300 affected individuals and their family/household members along with their data and specimens.

Data/Specimen Collection Procedures and Frequency: The only required study procedure is the review of medical records. Optional study procedures include collection of germline DNA (via blood, saliva, urine, or hair), plasma collection, stool collection, and skin biopsies. Clinical data will be updated every 6 months. Subjects can opt-out of this follow-up process.

ELIGIBILITY:
Inclusion Criteria:

Affected Patient (Group 1)

1. Males or females aged 0 and above.
2. Confirmed germline TP53 mutation or variant. OR Family history of LFS and clinically managed as a LFS patient. OR Meet LFS diagnostic criteria including Classic, Chompret, and LFL (Birch and Eeles) criteria.
3. Informed consent for capable participants. OR Parental/legally authorized representative permission (informed consent) for pediatric participants or subjects with diminished capacity, and if appropriate, assent.

Unaffected Family Member (Group 2)

1. Males or females aged 0 and above.
2. Biological relative of subjects with germline TP53 mutation or variant (LFS), including first degree (siblings, parents) and second degree (grandparents, aunts, uncles) relatives.
3. Negative for germline TP53 mutation or variant.
4. Informed consent for capable participants. OR Parental/legally authorized representative permission (informed consent) for pediatric participants or subjects with diminished capacity, and if appropriate, assent.

Household Member (Group 3)

1. Males or females aged 0 and above.
2. Household member of subjects with germline TP53 mutation or variant (LFS), sharing a living space (apartment or free-standing home) for at least 6 months prior to study enrollment.
3. Informed consent for capable participants. OR Parental/legally authorized representative (LAR) permission (informed consent) for pediatric participants or subjects with diminished capacity, and if appropriate, assent.

Exclusion Criteria:

1. Parents/LAR or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
2. Known pregnancy at the time of study enrollment.

Subjects that do not meet all of the enrollment criteria may not be enrolled. Pregnant women will not be actively enrolled, but if a woman becomes pregnant she will not be removed from the study; sample collection will be held during known pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with LFS/ LFL, family members, and household members
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2029-09-24 (Estimated); Study Completion 2029-09-24 (Estimated)

PRIMARY OUTCOMES:
Descriptive clinical data of all patients with confirmed germline TP53 variants | Five years
  These data include but are not limited to family history, cancer history, genetic testing, and cancer treatment.
Genomic landscape of TP53-associated tumors | Five years
Sequencing data from prospective blood collection and detection of ctDNA in plasma | Five years

SECONDARY OUTCOMES:
Utility of ctDNA assay in detection of cancer development in LFS patients | Five years
Genotype-phenotype correlations in patients with inherited TP53 mutations | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Kara N Maxwell, MD, PhD, Principal Investigator — University of Pennsylvania; Suzanne MacFarland, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Phildelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Only a limited data set will be available to future users of the biobank. To access data and biospecimens within the biobank, the prospective recipient executes a written Data User Agreement with the biobank, which will prohibit any attempts to re-identify subjects. Limited data will then be transmitted to prospective researchers using downloaded Excel compatible file formats. PHI will be maintained within the database as part of the consent process, in a partitioned and protected fashion (not available to future investigators) to permit the addition of updated clinical information into the biobank on a periodic basis. If for any reason the study is terminated, all data will be retained for six years, per CHOP policy A-3-9 for data retention. Following the end of data retention, data will be permanently de-coded and de-identified.